CLINICAL TRIAL: NCT03827018
Title: A Phase 2, Randomized, Double-blind Placebo-controlled Study to Test the Efficacy and Safety of KPL-301 in Giant Cell Arteritis
Brief Title: KPL-301 for Subjects With Giant Cell Arteritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kiniksa Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kiniksa Pharmaceuticals International, plc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPL-301-C001
Record Dates: First submitted 2019-01-25; First posted 2019-02-01 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Giant Cell Arteritis
Keywords: GCA; temporal arteritis; Horton's disease
MeSH Terms: conditions — Giant Cell Arteritis | interventions — mavrilimumab; Prednisone

STUDY DESIGN:
Intervention Model Description: Upon successful completion of the screening procedures, diagnosis criteria will be entered into an interactive web response system, and eligible subjects will be stratified for randomized study treatment into two cohorts according to whether subjects have new-onset or relapsing/refractory disease.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- mavrilimumab (Active Comparator): Subjects randomized to mavrilimumab will receive 150 mg every other week by subcutaneous injection co-administered with a 26-week corticosteroid taper.
  Interventions: Combination Product: mavrilimumab; Drug: prednisone
- placebo (Placebo Comparator): Subjects randomized to placebo will receive placebo every other week by subcutaneous injection co-administered with a 26-week corticosteroid taper.
  Interventions: Combination Product: placebo; Drug: prednisone

INTERVENTIONS:
Combination Product: mavrilimumab — 1 mL of 150 mg in a pre-filled syringe
  Other Names: KPL-301
  Arms: mavrilimumab
Combination Product: placebo — 1 mL of placebo in a pre-filled syringe
  Arms: placebo
Drug: prednisone — Prednisone tablets for oral administration containing either 1 mg, 2.5 mg, 5 mg, 10 mg, 20 mg or 50 mg of prednisone United States Pharmacopeia (USP)

SUMMARY:
The primary objective of the study is to evaluate the efficacy of mavrilimumab (KPL-301) versus placebo, co-administered with a 26-week corticosteroid taper, for maintaining sustained remission for 26 weeks in subjects with new onset or relapsing/refractory giant cell arteritis (GCA).

DETAILED DESCRIPTION:
This Phase 2 randomized, double-blind, placebo-controlled proof of concept study will evaluate the efficacy and safety of mavrilimumab co-administered with a 26-week corticosteroid taper in subjects with GCA. The study will consist of a screening period (up to 6 weeks), a 26-week double-blind placebo-controlled period during which subjects will receive blinded mavrilimumab or placebo co-administered with a 26-week corticosteroid taper, and a 12-week washout safety follow-up period during which subjects will discontinue and wash off blinded mavrilimumab or placebo.

ELIGIBILITY:
Selected Inclusion Criteria:

1. Subjects with new-onset or relapsing/refractory GCA.
2. Westergren erythrocyte sedimentation rate > 30 mm/hour or c-reactive protein ≥ 1 mg/ dL.
3. Remission of GCA at or before Day 0.
4. Female subjects must be postmenopausal or permanently sterile following documented hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or tubal ligation or having a male partner with vasectomy as affirmed by the subject, or nonpregnant, nonlactating, and if sexually active having agreed to use a highly effective method of contraception.
5. Male subjects must have documented vasectomy or if sexually active must agree to use a highly effective method of contraception with their partners of childbearing potential.

Selected Exclusion Criteria:

1. Transplanted organs (except corneal transplant performed more than 3 months prior to randomization).
2. Concurrent enrollment in another interventional clinical study.
3. Treatment with non-biologic investigational drug therapy within 4 weeks or 5 half-lives of the study agent, whichever was longer, prior to screening.
4. Cell-depleting biological therapies within 12 months prior to Day 0, or noncell-depleting biological therapies within 8 weeks (or 5 half-lives, whichever is longer) prior to screening.
5. Treatment with alkylating agents within 12 weeks prior to screening.
6. Intramuscular, Intra-articular or IV corticosteroids within 4 weeks prior to screening.
7. Receipt of live (attenuated) vaccine within the 4 weeks before Day 0.
8. Treatment with hydroxychloroquine, cyclosporine A, azathioprine, cyclophosphamide, or mycophenolate mofetil (MMF) within 4 weeks of screening.
9. Female subjects who are pregnant, intending to become pregnant, or are breastfeeding.
10. Known history of allergy or reaction to any component of the mavrilimumab or placebo formulation or to any other biologic therapy or prednisone or any of its excipients.
11. Positive (or 2 indeterminate) QuantiFERON test results.
12. Clinically significant active infection or infection requiring hospitalization or IV antibiotics within 12 weeks before screening or opportunistic infection within 6 months before screening.
13. Chronic active hepatitis B infection.
14. Subjects at a high risk of infection, a history of an infected joint prosthesis still in situ, leg ulcers, indwelling urinary catheter, or persistent or recurrent chest infections.
15. History of cancer within the last 10 years, except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured.
16. Evidence of clinically-uncontrolled respiratory disease.
17. History of chronic respiratory tract infections.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Paolini, M.D., Study Director — Kiniksa Pharmaceuticals, Ltd.
Locations (49):
- United States (8):
  - Site 1703, Sarasota, Florida
  - Site 1708, Tampa, Florida
  - Site 1706, Atlanta, Georgia
  - Site 1701, Boston, Massachusetts
  - Site 1707, Lansing, Michigan
  - Site 1704, Saint Clair Shores, Michigan
  - Site 1702, Rochester, Minnesota
  - Site 1705, New York, New York
- Australia (5):
  - Site 2102, Kogarah
  - Site 2105, Nedlands
  - Site 2106, Parkville
  - Site 2101, Victoria Park
  - Site 2104, Woodville South
- Belgium (4):
  - Site 2204, Brussels
  - Site 2202, Leuven
  - Site 2201, Liège
  - Site 2203, Yvoir
- Site 2303, Zagreb, Croatia
- Estonia (2):
  - Site 2401, Tallinn
  - Site 2402, Tartu
- Germany (7):
  - Site 2502, Tübingen, Baden-Wurttemberg
  - Site 2504, Erlangen, Bavaria
  - Site 2507, Freiburg im Breisgau
  - Site 2506, Hamburg
  - Site 2503, Hanover
  - Site 2508, Jena
  - Site 2501, Kirchheim unter Teck
- Site 2601, Dublin, Ireland
- Italy (4):
  - Site 2703, Milan
  - Site 2701, Pieve Emanuele
  - Site 2702, Reggio Emilia
  - Site 2704, Udine
- Netherlands (2):
  - Site 2802, Groningen
  - Site 2801, Rotterdam
- New Zealand (2):
  - Site 2902, Christchurch
  - Site 2901, Wellington
- Site 1002, Krakow, Poland
- Serbia (3):
  - Site 1101, Belgrade
  - Site 1102, Belgrade
  - Site 1103, Belgrade
- Site 1201, Ljubljana, Slovenia
- Spain (4):
  - Site 1303, A Coruña
  - Site 1301, Barcelona
  - Site 1304, Bilbao
  - Site 1302, Santa Cruz de Tenerife
- United Kingdom (4):
  - Site 1604, Edinburgh
  - Site 1603, Essex
  - Site 1602, London
  - Site 1601, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cid MC, Unizony SH, Blockmans D, Brouwer E, Dagna L, Dasgupta B, Hellmich B, Molloy E, Salvarani C, Trapnell BC, Warrington KJ, Wicks I, Samant M, Zhou T, Pupim L, Paolini JF; KPL-301-C001 Investigators. Efficacy and safety of mavrilimumab in giant cell arteritis: a phase 2, randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2022 May;81(5):653-661. doi: 10.1136/annrheumdis-2021-221865. Epub 2022 Mar 9. PMID 35264321

RESULTS

PARTICIPANT FLOW:
Groups:
- Mavrilimumab: Participants randomized to mavrilimumab receive 150 mg every other week by subcutaneous injection co-administered with a 26-week corticosteroid taper.
- Placebo: Participants randomized to placebo receive placebo every other week by subcutaneous injection co-administered with a 26-week corticosteroid taper.
Period: Overall Study
Arm/Group | Mavrilimumab | Placebo
Started | 42 | 28
Completed Treatment | 31 | 12
Completed (Completed Study) | 39 | 25
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mavrilimumab | Placebo | Total
Number analyzed (Participants) | 42 | 28 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (6.98) | 69.7 (8.31) | 69.7 (7.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 18 | 50
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 28 | 68
  Other, Not Specified | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 41 | 26 | 67

OUTCOME MEASURES:

1. Primary Outcome: Time to Flare by Week 26
Description: Time to flare by Week 26 was defined as time from randomization to the date of first flare occurring within the 26-week period, as assessed by independent adjudication. Kaplan-Meier method used to estimate the survival functions for each treatment arm.
  Flare/relapse was defined as a C-reactive protein (CRP) of 1 mg/dL or greater and/or erythrocyte sedimentation rate (ESR) of 30 mm/h or greater AND at least one of the following signs or symptoms attributed to GCA: Cranial symptoms (new-onset localized headache; scalp or temporal artery tenderness; ischemic-related vision loss; unexplained mouth or jaw pain upon mastication; transient ischemic attack or stroke related to GCA); Extracranial symptoms (claudication of the extremities; symptoms of polymyalgia rheumatica); New or worsening angiographic abnormalities detected via MRI, CT/CTA, or PET-CT of the aorta or other great vessels or via ultrasound of the temporal arteries.
Time Frame: Week 26
Population: Modified Intent to Treat (mITT) Analysis Set: all randomized participants who received at least 1 dose of mavrilimumab or placebo and had at least 1 assessment in the double-blind treatment period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 42 | 28
weeks | NA [NA to NA] — Not estimable per Kaplan-Meier method (insufficient number of subjects with events) | 25.1 [16.0 to NA] — Not estimable per Kaplan-Meier method (insufficient number of subjects with events)
Statistical Analysis 1: Comparison: Mavrilimumab vs Placebo; Test type: Superiority; p = 0.0263, Log Rank — Comparison of KPL-301 and placebo with respect to time to flare calculated by using a log-rank test stratified by randomization strata; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.15 to 0.92] — 95% confidence interval was calculated based on a Cox proportional-hazards model with treatment as covariate and stratified by randomization strata

2. Secondary Outcome: Sustained Remission Rate at Week 26
Description: The sustained remission rate at Week 26 is defined as the percentage of participants with sustained remission, as assessed by independent adjudication, at Week 26, derived from the time to flare curve. Kaplan-Meier Survival Estimates with standard error and 95% CI for each arm. Participants who completed the treatment period without a flare by Week 26 were considered to have sustained remission.
Time Frame: Week 26
Population: mITT Analysis Set: all randomized participants who received at least 1 dose of mavrilimumab or placebo and had at least 1 assessment in the double-blind treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 42 | 28
percentage of participants | 83.2 [67.9 to 91.6] | 49.9 [29.6 to 67.3]
Statistical Analysis 1: Comparison: Mavrilimumab vs Placebo; Secondary endpoints were analyzed in hierarchical order; Test type: Superiority; p = 0.0038, normal approximation — Two-sided p-value and 95% CI for the difference in sustained remission between two arms using normal approximation. Placebo arm is the reference; Difference in proportions = 33.3, 95% CI 2-sided [10.7 to 55.8]

3. Secondary Outcome: Time to Elevated Erythrocyte Sedimentation Rate (ESR) by Week 26
Description: Elevated ESR is defined as first occurrence of ESR value ≥ 30 mm/hr. Participants with elevated ESR within 3 days of first dose are excluded from the analysis. Kaplan-Meier method used to estimate the survival functions for each treatment arm.
Time Frame: Week 26
Population: mITT Analysis Set: all randomized participants who received at least 1 dose of mavrilimumab or placebo and had at least 1 assessment in the double-blind treatment period. Participants with elevated ESR within 3 days of first dose are excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 40 | 28
weeks | 26.1 [16.1 to NA] — Not estimable per Kaplan-Meier method (insufficient number of subjects with events) | 12.1 [8.1 to 16.6]
Statistical Analysis 1: Comparison: Mavrilimumab vs Placebo; Secondary endpoints were analyzed in hierarchical order; Test type: Superiority; p = 0.0277, Log Rank — Calculated by using a log-rank test stratified by randomization strata; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.27 to 0.95] — Calculated based on a Cox proportional-hazards model with treatment as covariate, and stratified by randomization strata

4. Secondary Outcome: Time to Elevated C-Reactive Protein (CRP) by Week 26
Description: Elevated CRP is defined as first occurrence of CRP value ≥ 1.0 mg/dL. Participants with elevated CRP within 3 days of first dose are excluded from the analysis. Kaplan-Meier method used to estimate the survival functions for each treatment arm.
Time Frame: Week 26
Population: mITT Analysis Set: all randomized participants who received at least 1 dose of mavrilimumab or placebo and had at least 1 assessment in the double-blind treatment period. Participants with elevated CRP within 3 days of first dose are excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 39 | 27
weeks | NA [8.1 to NA] — Not estimable per Kaplan-Meier method (insufficient number of subjects with events) | 12.3 [3.3 to 24.1]
Statistical Analysis 1: Comparison: Mavrilimumab vs Placebo; Secondary endpoints were analyzed in hierarchical order; Test type: Superiority; p = 0.0378, Log Rank — Calculated by using a log-rank test stratified by randomization strata; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.19 to 0.98] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Time to Signs/Symptoms of Giant Cell Arteritis (GCA) or New or Worsening Vasculitis on Imaging by Week 26
Description: Kaplan-Meier method used to estimate the survival functions for each treatment arm.
Time Frame: Week 26
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 42 | 28
weeks | NA [NA to NA] — Not estimable per Kaplan-Meier method (insufficient number of subjects with events) | 25.1 [15.1 to NA] — Not estimable per Kaplan-Meier method (insufficient number of subjects with events)
Statistical Analysis 1: Comparison: Mavrilimumab vs Placebo; Secondary endpoints were analyzed in hierarchical order; Test type: Superiority; p = 0.0651, Log Rank — Calculated by using a log-rank test stratified by randomization strata; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.22 to 1.06] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Cumulative Corticosteroid Dose at Week 26
Time Frame: Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 42 | 28
mg | 2074.15 (708.433) | 2402.98 (1014.446)
Statistical Analysis 1: Comparison: Mavrilimumab vs Placebo; Test type: Other — Descriptive statistic; p = 0.0667, ANCOVA — Calculated using ANCOVA with treatment arm and randomization strata as discrete variables, and corticosteroid starting dose as a continuous variable; Least Squares (LS) means difference = -326.45, 95% CI 2-sided [-675.99 to 23.09]

7. Secondary Outcome: Percentage of Participants Who Completed the 26-Week Corticosteroid Taper and Who Had a Normal ESR
Description: Participants were considered to have completed the corticosteroid taper if by week 26 receiving 1 mg/day for those who start with 60 mg/day, or 0 mg/day for those who start with doses < 60 mg/day. 95% CI calculated using Clopper-Pearson confidence intervals.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 42 | 28
percentage of participants | 45.2 [29.8 to 61.3] | 14.3 [4.0 to 32.7]
Statistical Analysis 1: Comparison: Mavrilimumab vs Placebo; Test type: Other — Descriptive statistic; p = 0.0201, Cochran-Mantel-Haenszel — 95% CI and p-value are analyzed using a Cochran-Mantel-Haenszel (CMH) test stratified by randomization strata; Difference in percentages = 31.0, 95% CI 2-sided [11.1 to 50.8]

8. Secondary Outcome: Percentage of Participants Who Completed the 26-Week Corticosteroid Taper and Who Had a Normal CRP Level
Description: as for outcome 7
Time Frame: Week 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 42 | 28
percentage of participants | 23.8 [12.1 to 39.5] | 14.3 [4.0 to 32.7]
Statistical Analysis 1: Comparison: Mavrilimumab vs Placebo; Test type: Other — Descriptive statistic; p = 0.5533, Cochran-Mantel-Haenszel — 95% CI and p-value are analyzed using a Cochran-Mantel-Haenszel (CMH) test stratified by randomization strata; Difference in percentages = 9.5, 95% CI 2-sided [-8.7 to 27.8]

9. Secondary Outcome: Percentage of Participants Who Completed the 26-week Corticosteroid Taper and Who Had No Signs or Symptoms of GCA Nor New or Worsening Vasculitis by Imaging by Week 26
Description: as for outcome 7
Time Frame: Week 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 42 | 28
percentage of participants | 71.4 [55.4 to 84.3] | 32.1 [15.9 to 52.4]
Statistical Analysis 1: Comparison: Mavrilimumab vs Placebo; Test type: Other — Descriptive statistics; p = 0.0031, Cochran-Mantel-Haenszel — 95% CI and p-value are analyzed using a Cochran-Mantel-Haenszel (CMH) test stratified by randomization strata; Difference in percentages = 39.3, 95% CI 2-sided [17.2 to 61.3]

10. Secondary Outcome: Cumulative Corticosteroid Dose at the End of the Washout Safety Follow-up Period
Time Frame: Final Safety Follow-up visit (Week 38)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 42 | 28
mg | 2464.93 (1106.636) | 2845.45 (1320.115)
Statistical Analysis 1: Comparison: Mavrilimumab vs Placebo; Test type: Other — Descriptive statistics; p = 0.1629, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares (LS) means difference = -380.82, 95% CI 2-sided [-919.66 to 158.02]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From signing of informed consent (up to 6 weeks prior to Baseline) through Final Safety Follow-up / Week 38 Adverse Events: from first dose of study drug through Final Safety Follow-up / Week 38
Arm/Group | Mavrilimumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/42 | 3/28
Other Adverse Events (participants affected / at risk) | 33/42 | 25/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mavrilimumab (N=42) | Placebo (N=28)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mavrilimumab (N=42) | Placebo (N=28)
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2
Oedema peripheral (General disorders) | 2 | 2
Pyrexia (General disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 5 | 3
Oral herpes (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 5
Carbon monoxide diffusing capacity decreased (Investigations) | 4 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 6 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 2
Sleep disorder (Psychiatric disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the sole and exclusive right to publish information obtained from the trial. PI has no right to publish. PI may be invited to publish.

DOCUMENTS (2):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT03827018/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT03827018/SAP_001.pdf